CLINICAL TRIAL: NCT04587791
Title: Cannabidiol Pharmacotherapy for Co-occurring Opioid Use Disorder and Chronic Pain
Brief Title: Cannabidiol in Opioid Use Disorder and Chronic Pain
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joao De Aquino, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JD001; 2000029286 (Other: Yale HRPP); 1K23DA052682-01 (NIH)
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Opioid Use Disorder
Keywords: Methadone; Buprenorphine; Cannabidiol; Pain
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Pain | interventions — Cannabidiol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: participants will receive CBD (400 mg, 800 mg, 1200 mg) or placebo.
Who Masked: Participant, Investigator
Masking Description: participants will receive CBD (400 mg, 800 mg, 1200 mg) or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CBD 400mg (Active Comparator): CBD 400 mg
  Interventions: Drug: 400mg Cannabidiol
- CBD 800mg (Active Comparator): CBD 800mg
  Interventions: Drug: 800mg Cannabidiol
- CBD 1200mg (Active Comparator): CBD 1200mg
  Interventions: Drug: 1200mg Cannabidiol
- Saline (Placebo Comparator): saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 400mg Cannabidiol — Participants will receive 400mg
  Other Names: CBD
  Arms: CBD 400mg
Drug: 800mg Cannabidiol — Participants will receive 800mg
  Other Names: CBD
  Arms: CBD 800mg
Drug: 1200mg Cannabidiol — Participants will receive 1200mg
  Other Names: CBD
  Arms: CBD 1200mg
Drug: Saline — Participants will receive saline
  Other Names: placebo
  Arms: Saline

SUMMARY:
This is a double-blind, randomized, placebo-controlled cross-over human laboratory study with a duration of approximately 4 weeks, during which participants will come to the testing site for a total of five times: one initial screening session, and four experimental sessions where study medication, Cannabidiol (CBD) will be administered, separated by at least 72 hours to limit carryover effects.

DETAILED DESCRIPTION:
Thirty-six male and female (ages 18-70) participants with comorbid opioid use disorder (OUD) and non-cancer chronic pain for at least 6 months, currently receiving methadone (n= 22) or buprenorphine (n= 12), will be enrolled. Prior to their daily methadone or buprenorphine dose and thus at trough plasma levels of opioid, participants will receive oral CBD (400 mg, 800 mg, 1200 mg) or placebo. Subsequently, all participants will undergo laboratory testing of opioid-related outcomes.

Pain sensitivity will be measures including the well-validated, Quantitative Sensory Testing (QST), the Pain Catastrophizing Scale (PCS), and a pain Visual Analog Scale (VAS). Attentional bias and cue-induced opioid craving will be measured using a visual probe task and the Heroin Craving Scale (HCQ-14). Abuse potential will be measured using the Drug Effects Questionnaire (DEQ). Negative affect will be measured using the Positive and Negative Affect Schedule (PANAS). Cognitive performance will be measured by a comprehensive cognitive battery that includes the Continuous Performance Test (CPT) and the Hopkins Verbal Learning Test (HVLT). Safety will be thoroughly measured with the Systematic Assessment for Treatment Emergent Events (SAFTEE) for adverse effects.

The order of study medication administration will be counterbalanced order to minimize carryover effects. On the initial screening day and at the end of medication treatment, blood will be drawn to determine serum drug levels. Participants will be thoroughly evaluated by a physician prior to discharge on each experimental session. One week after the last study medication dose, participants will be conducted by phone for a follow-up session.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, Veterans and non-Veterans, aged between 18 and 70 years old.
* Diagnosed with OUD and currently enrolled in methadone or buprenorphine maintenance treatment.
* Having chronic pain, uniformly operationalized as grade II (high-intensity) non-cancer musculoskeletal pain for ≥ 6 months 49
* Capable of providing informed consent in English.
* Compliant in opioid maintenance treatment and on a stable dose for two weeks or longer.
* Not meeting DSM-5 criteria for substance use disorders other than OUD or tobacco use disorder within the last 12 months.
* No current medical problems deemed contraindicated for participation by principal investigator.
* For women, not pregnant as determined by pregnancy screening; not breast-feeding; using acceptable birth control methods.

Exclusion Criteria:

* Other current major psychiatric disorders deemed clinically unstable by the principal investigator, such as severe depression and/or active suicidal ideation.
* Having experienced major psychosocial stressors recently (≤ 6 weeks before enrollment), at the discretion of the principal investigator.
* Having received inpatient psychiatric treatment recently (≤ 60 days before enrollment).
* A study physician will determine if participants receiving products containing THC or CBD products may participate in the study.
* Current use benzodiazepines or platelet inhibitors (e.g., clopidogrel, apixaban, ticagrelor).
* Current weight of less of 60 kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Variable #1: Safety and tolerability of CBD | Baseline and up to 6 hours
  To monitor adverse events from the study medications, the Systematic Assessment for Treatment Emergent Events (SAFTEE) will be administered before and after each experimental session. This is a symptom checklist that has been used successfully in our previous studies to assess possible side effects of study medications. It includes information regarding severity of any presenting side effects, as well as the course of action taken by study staff in response.
Primary Outcome Variable #2: Pain Sensitivity | Baseline and up to 6 hours
  We will measure pain sensitivity using a comprehensive QST battery at baseline and approximately hourly for 6 hours.
Primary Outcome Variable #3: Abuse potential of CBD (DEQ) | Baseline and up to 6 hours
  The abuse potential of CBD will be assessed using the Drug Effects Questionnaire (DEQ) administered at baseline and every 30 minutes. The primary DEQ outcome is the Stimulatory Effects subscale, obtained by averaging participants responses to the items: "Feel High"; "Feel Stimulated"; and "Feel the Drug Strength".
Primary Outcome Variable #4A: Cognitive/psychomotor effects (CPT) | +210 minutes post dose
  The cognitive/psychomotor effects of CBD will be assessed using the Continuous Performance Test (CPT). For the CPT, the primary outcome will be the throughput score, which indexes attention/working memory accuracy (i.e. percent of correct responses) and speed (i.e. reaction time).
Primary Outcome Variable #4B: Cognitive/psychomotor effects (HVLT) | +210 minutes post dose
  The cognitive/psychomotor effects of CBD will be assessed using the Hopkins Verbal Learning Test (HVLT). The primary outcome for the HVLT will be immediate and delayed recall, which index verbal memory.

SECONDARY OUTCOMES:
Secondary Outcome Variable #1: Opioid Craving | Baseline and +150 minutes post dose
  We will measure opioid craving using the short form Heroin Craving Questionnaire (HCQ-14) given to participants before and after a watching a visual probe task used to induce craving.

OTHER OUTCOMES:
Influence of sex | Up to 6 hours
  We will explore if sex moderates the relationships hypothesized in the primary and secondary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Joao De Aquino, M.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs Hospital, West Haven, Connecticut, United States